CLINICAL TRIAL: NCT02387164
Title: Double-blind, Investigator-initiated Study to Determine the Effect of Alum-GAD (Diamyd) in Combination With Vitamin D3 on the Progression to Type 1 Diabetes in Children With Multiple Islet Autoantibodies
Brief Title: Prevention Trial: Immune-tolerance With Alum-GAD (Diamyd) and Vitamin D3 to Children With Multiple Islet Autoantibodies
Acronym: DiAPREV-IT2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was interrupted early and terminated when only 26 out of 80 patients were enrolled due to new clinical study results indicating that the current study would not be informative.
Sponsor: Lund University (Other)
Collaborators: Region Skane (Other)
Responsible Party: Principal Investigator, Helena Elding Larsson, Docent, MD, PhD, Lund University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DiAPREV/2014
Record Dates: First submitted 2015-03-05; First posted 2015-03-12 (Estimated); Results first posted 2020-10-27 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus, Type 1; Prediabetic State
Keywords: Type 1 diabetes; Islet autoantibodies; glutamate decarboxylase autoantibodies (GADA); Immune tolerance; Prediabetes; Glucose tolerance; glutamate decarboxylase; Prevention; Children
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Prediabetic State | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alum-GAD, Vitamin D3 (Experimental): Two doses à 20 microgram of subcutaneous alum-GAD (Diamyd), 30 Days apart. Vitamin D 2000 U/Daily with start 30 days before the first injection of Diamyd. Vitamin D treatment will continue throughout the whole study period of 5 years.
  Interventions: Drug: Alum-GAD; Drug: Vitamin D3
- Placebo, Vitamin D3 (Placebo Comparator): Two doses of subcutaneous placebo, 30 Days apart. Vitamin D 2000 U/Daily with start 30 days before the first injection of Diamyd. Vitamin D treatment will continue throughout the whole study period of 5 years
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Alum-GAD — Two doses à 20 microgram 30 days apart subcutaneously administrated
  Other Names: Diamyd; GAD-Alum; Alumformulated GAD
  Arms: Alum-GAD, Vitamin D3
Drug: Vitamin D3 — 2000 Units (IE) (50 microgram) vitamin D3 daily
  Other Names: Cholecalciferol

SUMMARY:
The purpose of this study is to evaluate if immune-tolerance with Alum-formulated GAD (Diamyd), in combination with high dose Vitamin D3, may delay or stop the autoimmune process leading to clinical type 1 diabetes in non-diabetic children with ongoing beta-cell autoimmunity as indicated by positive islet autoantibodies.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate if immune-tolerance with Alum-formulated GAD (Diamyd), combined with high dose Vitamin D3, may delay or stop the autoimmune process leading to clinical type 1 diabetes (diagnosed according to American Diabetes Association criteria) in non-diabetic 4-17.99 year old children with ongoing beta-cell autoimmunity as indicated by positive islet autoantibodies.

The secondary objective is to demonstrate that treatment with Diamyd is safe in children at risk for type 1 diabetes.

The children will be followed for 5 years in the study. Primary endpoint is proportion of subjects diagnosed with type 1 diabetes in each treatment arm. Secondary endpoints are 1) safety, 2) change in metabolic status from normal to impaired glucose metabolism in the group of children with normal glucose metabolism at baseline screening.

ELIGIBILITY:
Inclusion Criteria:

* Children 4-17.99 years of age with positive autoantibodies to glutamate decarboxylase (GADA) and at least one additional type 1 diabetes associated autoantibody (to insulinoma associated protein 2 (IA-2A), Zinktransporter 8 (ZnT8R/Q/WA) or insulin (IAA)).
* Written informed consent from the child and the childs legal representative(s).

Exclusion Criteria:

1. Ongoing treatment with immunosuppressant therapy.
2. Diabetes.
3. Treatment with any oral or injected anti-diabetic medications
4. Significantly abnormal hematology results at screening.
5. Clinically significant history of acute reaction to vaccines or other drugs
6. Treatment with any vaccine within one month prior to the first dose of the study drug or planned treatment with vaccine up to three months after the last injection with the study drug.
7. A history of epilepsy, serious head trauma or cerebrovascular accident, or Clinical features of continuous motor unit activity in proximal muscles
8. Participation in other Clinical trials with a new chemical entity within the previous 3 months.
9. History of hypercalcemia.
10. Unwilling to abstain from other medication with Vitamin D during the study period.
11. Significant illness within 2 weeks prior to first dosing.
12. Known Human Immuno Deficiency Virus infection or hepatitis.
13. Presence of associated serious disease or condition.
14. Diabetes-protective Human Leucocyte Antigen (HLA) DQ6.
15. Females who are lactating or pregnant.
16. Males or females not willing to use adequate contraception, if sexually active, until 1 year after the last Diamyd administration.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2015-03-09 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2019-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helena Elding Larsson, MD, PhD, Principal Investigator — Lund University
Locations (1):
- Clinical Research Center, Pediatric Endocrinology, Jan Waldenströms gata 35, 60:11, Malmo, Sweden

REFERENCES:
- [Background] Elding Larsson H, Larsson C, Lernmark A; DiAPREV-IT study group. Baseline heterogeneity in glucose metabolism marks the risk for type 1 diabetes and complicates secondary prevention. Acta Diabetol. 2015 Jun;52(3):473-81. doi: 10.1007/s00592-014-0680-1. Epub 2014 Nov 8. PMID 25381193
- [Background] Andersson C, Carlsson A, Cilio C, Cedervall E, Ivarsson SA, Jonsdottir B, Jonsson B, Larsson K, Neiderud J, Lernmark A, Elding Larsson H; DiAPREV-IT Study Group. Glucose tolerance and beta-cell function in islet autoantibody-positive children recruited to a secondary prevention study. Pediatr Diabetes. 2013 Aug;14(5):341-9. doi: 10.1111/pedi.12023. Epub 2013 Mar 8. PMID 23469940
- [Background] Ludvigsson J, Krisky D, Casas R, Battelino T, Castano L, Greening J, Kordonouri O, Otonkoski T, Pozzilli P, Robert JJ, Veeze HJ, Palmer J, Samuelsson U, Elding Larsson H, Aman J, Kardell G, Neiderud Helsingborg J, Lundstrom G, Albinsson E, Carlsson A, Nordvall M, Fors H, Arvidsson CG, Edvardson S, Hanas R, Larsson K, Rathsman B, Forsgren H, Desaix H, Forsander G, Nilsson NO, Akesson CG, Keskinen P, Veijola R, Talvitie T, Raile K, Kapellen T, Burger W, Neu A, Engelsberger I, Heidtmann B, Bechtold S, Leslie D, Chiarelli F, Cicognani A, Chiumello G, Cerutti F, Zuccotti GV, Gomez Gila A, Rica I, Barrio R, Clemente M, Lopez Garcia MJ, Rodriguez M, Gonzalez I, Lopez JP, Oyarzabal M, Reeser HM, Nuboer R, Stouthart P, Bratina N, Bratanic N, de Kerdanet M, Weill J, Ser N, Barat P, Bertrand AM, Carel JC, Reynaud R, Coutant R, Baron S. GAD65 antigen therapy in recently diagnosed type 1 diabetes mellitus. N Engl J Med. 2012 Feb 2;366(5):433-42. doi: 10.1056/NEJMoa1107096. PMID 22296077
- See also: Link to the description of the first DiAPREV-IT study, that have included 50 children and is still ongoing — http://www.ludc.med.lu.se/research-units/diabetes-and-celiac-disease/research-projects/diabetes-prevention-immune-tolerance/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 29 patients were screened for the study and 26 entered the study. Three patients were screening failures.
Groups:
- Alum-GAD, Vitamin D3: Two doses à 20 microgram of subcutaneous alum-GAD (Diamyd), 30 Days apart. Vitamin D 2000 U/Daily with start 30 days before the first injection of Diamyd. Vitamin D treatment will continue throughout the whole study period of 5 years.
  Alum-GAD (Glutamic Acid Decarboxylase): Two doses à 20 microgram 30 days apart subcutaneously administrated
  Vitamin D3: 2000 Units (IE) (50 microgram) vitamin D3 daily
Period: Overall Study
Arm/Group | Alum-GAD, Vitamin D3 | Placebo, Vitamin D3
Started | 13 | 13
Completed | 10 | 11
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Diagnosed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alum-GAD, Vitamin D3 | Placebo, Vitamin D3 | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 13 | 26
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.0 (2.89) | 9.4 (2.73) | 9.2 (2.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 6 | 9 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 13 | 13 | 26
Weight [Mean (Standard Deviation); unit: kg] | 33.7 (14.51) | 36.6 (14.99) | 35.1 (14.53)
Celiac disease [Count of Participants; unit: Participants]
  Yes | 2 | 0 | 2
  No | 11 | 13 | 24
Thyroid disease [Count of Participants; unit: Participants]
  Yes | 0 | 0 | 0
  No | 13 | 13 | 26
Relatedness [Count of Participants; unit: Participants]
  First degree relative diagnosed with type 1 diabetes | 4 | 2 | 6
  General population (no relative diagnosed with type 1 diabetes) | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Type 1 Diabetes Month 24
Description: Number of patients diagnosed with type 1 diabetes according to ADA (American Diabetes Association) criteria in each study arm month 24
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Alum-GAD, Vitamin D3 | Placebo, Vitamin D3
Number analyzed (Participants) | 13 | 13
Participants
  Yes | 1 | 2
  No | 12 | 11

2. Primary Outcome: Type 1 Diabetes Status Overall
Description: Number of patients diagnosed with type 1 diabetes according to ADA (American Diabetes Association) criteria in each study arm overall. Including one patient diagnosed shortly after the month 24 visit.
Time Frame: Over the entire study period up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Alum-GAD, Vitamin D3 | Placebo, Vitamin D3
Number analyzed (Participants) | 13 | 13
Participants
  Yes | 2 | 2
  No | 11 | 11

3. Secondary Outcome: Number of Patients Developing Impaired Glucose Metabolism Until Month 18
Description: Change in metabolic status from normal to impaired glucose metabolism during follow-up in the group of children with normal glucose metabolism at baseline screening.
  Impaired glucose metabolism is defined as a) fasting plasma glucose 6.1 mmol/L or more, b) maximum plasma glucose 30, 60, 90 min during oral glucose tolerance test (OGTT) 11.1 mmol/L or more, c) 120 min plasma glucose on OGTT 7.8 mmol/L or more, d) HbA1c 39 mmol/L or more.
Time Frame: During 18 months follow-up
Population: Only patients with normal glucose at baseline and glucose measured at month 18 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Alum-GAD, Vitamin D3 | Placebo, Vitamin D3
Number analyzed (Participants) | 8 | 6
Participants
  Yes | 3 | 1
  No | 5 | 5

4. Secondary Outcome: Number of Patients With Progressive Impaired Glucose Metabolism Until Month 18
Description: Number of patients who have progression from already impaired glucose metabolism from one or several criteria to additional signs of reduced glucose metabolism (within children with impaired glucose metabolism at screening).
  Impaired glucose metabolism is defined as a) fasting plasma glucose 6.1 mmol/L or more, b) maximum plasma glucose 30, 60, 90 min during oral glucose tolerance test (OGTT) 11.1 mmol/L or more, c) 120 min plasma glucose on OGTT 7.8 mmol/L or more, d) HbA1c 39 mmol/L or more.
Time Frame: During 18 months follow-up
Population: Only patients with impaired glucose at baseline and glucose measured at month 18 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Alum-GAD, Vitamin D3 | Placebo, Vitamin D3
Number analyzed (Participants) | 2 | 4
Participants
  Yes | 1 | 0
  No | 1 | 4

5. Secondary Outcome: Injection Site Reactions Day 1
Description: Number of patients experiencing injection site reactions at day 1
Time Frame: Day 1
Measure: Number; unit: participants
Arm/Group | Alum-GAD, Vitamin D3 | Placebo, Vitamin D3
Number analyzed (Participants) | 13 | 13
participants
  Erythema | 0 | 0
  Haematoma | 0 | 0
  Itching | 0 | 0
  Oedema | 0 | 0
  Pain | 0 | 0
  Tenderness | 0 | 0

6. Secondary Outcome: Injection Site Reactions Month 1
Description: Number of patients experiencing injection site reactions at month 1
Time Frame: Month 1
Measure: Number; unit: participants
Arm/Group | Alum-GAD, Vitamin D3 | Placebo, Vitamin D3
Number analyzed (Participants) | 13 | 13
participants
  Erythema | 1 | 0
  Haematoma | 1 | 0
  Itching | 0 | 0
  Oedema | 2 | 0
  Pain | 0 | 0
  Tenderness | 0 | 0

7. Secondary Outcome: Change From Baseline in GADA Month 1
Description: Change from baseline to month 1 in GADA (Glutamic Acid Decarboxylase Antibodies) titers
Time Frame: Month 1
Population: Only patients with GADA measured both at baseline and month 1 are included.
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Alum-GAD, Vitamin D3 | Placebo, Vitamin D3
Number analyzed (Participants) | 13 | 12
U/mL | 1619.1 (2608.9) | -51.9 (197.8)

8. Secondary Outcome: Change From Baseline in GADA Month 12
Description: Change from baseline to month 12 in GADA titers
Time Frame: Month 12
Population: Only patients with GADA measured at baseline and at month 12 are included.
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Alum-GAD, Vitamin D3 | Placebo, Vitamin D3
Number analyzed (Participants) | 10 | 10
U/mL | 7916.9 (10694.55) | -120.0 (592.09)

9. Secondary Outcome: Change From Baseline in GADA Month 24
Description: Change from baseline to month 24 in GADA titers
Time Frame: Month 24
Population: Only patients with GADA measured at baseline and month 24 are included.
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Alum-GAD, Vitamin D3 | Placebo, Vitamin D3
Number analyzed (Participants) | 9 | 11
U/mL | 3216.6 (4628.53) | 1062.7 (3380.26)

ADVERSE EVENTS:
Time Frame: During the entire study period approximately 24 months.
Description: At each study visit the investigator asked for any adverse events and recorded them in the CRF (Case Report Form).
Arm/Group | Alum-GAD, Vitamin D3 | Placebo, Vitamin D3
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/13 | 1/13
Other Adverse Events (participants affected / at risk) | 12/13 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alum-GAD, Vitamin D3 (N=13) | Placebo, Vitamin D3 (N=13)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post streptococcal glomerulonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alum-GAD, Vitamin D3 (N=13) | Placebo, Vitamin D3 (N=13)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (2)
Headache (Nervous system disorders) | 5 (13) | 3 (9)
Migraine (Nervous system disorders) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 4 (6) | 5 (11)
Pain (General disorders) | 2 (3) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Injection site rash (General disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (2) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 10 (49) | 9 (20)
Ear infection (Infections and infestations) | 3 (3) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3) | 1 (3)
Influenza (Infections and infestations) | 2 (3) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Enterobiasis (Infections and infestations) | 0 (0) | 1 (2)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Growing pains (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Attention deficit/hyperactivit (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was interrupted early and terminated when only 26 out of 80 patients were enrolled. The patients were followed for 2 years rather than the planned 5 years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/64/NCT02387164/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/64/NCT02387164/SAP_001.pdf